CLINICAL TRIAL: NCT01710007
Title: A Prospective, Double-blind, Randomized, Parallel, Multiple-center Study to Compare the Efficacy and Safety of 1PC002 and Atorvastatin in Taiwanese Patients With Hypercholesterolemia
Brief Title: Efficacy and Safety Study of Pitavastatin for Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QCR10022
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Hypercholesterolemia
Keywords: HMG-CoA reductase inhibitors
MeSH Terms: conditions — Hypercholesterolemia | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1PC002 (Experimental): 2 mg 1PC002 once daily for 12 weeks.
  Interventions: Drug: 1PC002
- Lipitor (Active Comparator): 10 mg atorvastatin once daily for 12 weeks.
  Interventions: Drug: Lipitor

INTERVENTIONS:
Drug: 1PC002 — Subjects should be instructed to take 1 capsule of study drug (1PC002 or atorvastatin) orally once a day, with or without food. Administration before bedtime or at regular time-interval is recommended.
  Other Names: Pitavastatin
  Arms: 1PC002
Drug: Lipitor — Subjects should be instructed to take 1 capsule of study drug (1PC002 or atorvastatin) orally once a day, with or without food. Administration before bedtime or at regular time-interval is recommended.
  Other Names: Atorvastatin
  Arms: Lipitor

SUMMARY:
1PC002 is a newly developed synthetic and highly potent HMG-CoA reductase inhibitor. Its active compound, pitavastatin has recently been approved by US FDA for indications of primary hypercholesterolemia and combined dyslipidaemia. It exhibits unique pharmacokinetic properties. Unlike atorvastatin which is metabolized by CYP3A4, metabolism of 1PC002 does not depend on CYP3A4. This multi-center study is conducted to confirm the efficacy and safety of 1PC002 administered for 12 weeks is non-inferior to atorvastatin.

DETAILED DESCRIPTION:
This is a prospective, active-controlled, double-blind, randomized, parallel, and multi-center study. To target 150 evaluable subjects, approximately 200 Taiwanese patients with primary hypercholesterolemia or combined dyslipidemia will be enrolled in this study.

After providing the written inform consent, patients will undergo a complete physical examination, vital sign (brachial BP / HR), medical history, and lab assessment, including fasting serum LDL-C, TC, HDL-C, TG, and non-HDL. They should not take any hypolipidemic drugs for at least 4 weeks prior to initiation of study treatment. All eligible subjects will be randomized into 2 groups in a 1:1 ratio to receive either 2 mg 1PC002 or 10 mg atorvastatin once daily for 12 weeks.

* Study Group: 1PC002 1 cap. q.d. p.o.
* Control Group: Atorvastatin 1 cap. q.d. p.o.

After entering the baseline visit, lipid profiles (including fasting serum LDL-C, TC, HDL-C, TG, non-HDL, Apo A1, Apo B and Apo B / Apo A1 ratio), hs-CRP, eGFR, spot urinary albumin / creatinine ratio (ACR) and central BP values will be obtained at baseline, Week 4 and Week 12 for evaluating the effectiveness of study drugs and for any possible changes in laboratory data. Non-HDL value will be calculated by subtracting HDL-C from TC. Moreover, serum Cystatin C, another biomarker of renal function, will also be assessed at baseline and Week 12.

For monitoring the safety, biochemical and hematological assessment will be performed at baseline, Week 4 and 12. Additional liver function and CK test will be conducted at Week 8. The occurring AE(s) and SAE will be followed until resolution or the event is considered stable.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males aged between 20 and 80 years.
2. Subjects who meet All of the following diagnosis at screening visit:

   * Primary hypercholesterolemia or combined dyslipidemia
   * TC ≥ 220 mg/dL or LDL-C ≥ 130 mg/dL
   * TG < 400 mg/dL
3. Subjects who is willing and able to provide ICF.

Exclusion Criteria:

1. Females who are pregnant, breast-feeding or intent to be pregnant during study period, or those of childbearing potential not using effective contraception.
2. Subject with documented homozygous familial hypercholesterolemia.
3. Subject with documented HIV.
4. Subject with documented hypothyroidism and inadequate treatment judged by investigator.
5. Subjects with unstable cardiovascular disease (CVD) prior to randomization.
6. Subjects with hepatic or biliary disorders, such as acute hepatitis, acute exacerbation of chronic hepatitis, liver cirrhosis, liver cancer and jaundice.
7. Any condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs.
8. Subjects with the following lab data at screening visit:

   * serum creatine kinase (CK) > 5 x upper limit of normal (ULN)
   * ALT or AST of > 3 x ULN
   * serum creatinine ≥ 1.5 mg/dL
   * HbA1c > 8.0%
9. Subject with the following past histories:

   * hypersensitivity to statins or any other ingredients of study drugs
   * resistant to statins treatment
10. Use of any lipid-lowering agents within 4 weeks prior to the initiation of study treatment.
11. Use of any investigational product within 4 weeks prior to screening.
12. Any unstable concomitant disease or clinical condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk to participate in the study or confounds the ability to interpret data from the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiau-Suong Liau, Principal Investigator — Buddhist Taipei TzuChi General Hospital; Ming-Shien Wen, Principal Investigator — Chang Gung Medical Foundation- LinKuo Branch; Wen-Pin Huang, Principal Investigator — Cheng-Hsin General Hospital; Dee Pei, Principal Investigator — Cardinal Tien Hospital; Wei-Shiang Lin, Principal Investigator — Tri-Service General Hospital; Huey-Herng Sheu, Principal Investigator — Taichung Veterans General Hospital; Chen-Huan Chen, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Ju-Chi Liu, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (8):
- Taiwan (8):
  - Buddhist Taipei TzuChi General Hospital, New Taipei City
  - Cardinal Tien Hospital, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation- LinKuo Branch, Taoyuan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1PC002 | Lipitor
Started | 103 | 99
Completed | 87 | 81
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1PC002 | Lipitor | Total
Number analyzed (Participants) | 103 | 99 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 93 | 180
  >=65 years | 16 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.36 (10.50) | 57.90 (8.80) | 56.60 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 57 | 117
  Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 103 | 99 | 202
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 103. | 99 | 202

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change From Baseline in LDL-C Level at Week 12.
Description: The study aimed to test that the efficacy of 1PC002 group was non-inferior to Atorvastatin group in percent change from baseline of LDL-C level at Week 12.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Lipitor | 1PC002
Number analyzed (Participants) | 94 | 100
Percent change from baseline | -42.89 (12.80) | -37.43 (17.97)

2. Secondary Outcome: LDL-C
Description: Percent change from baseline in LDL-C level at Week 4
Time Frame: week 4
Population: ITT population had been analysis
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | 1PC002 | Lipitor
Number analyzed (Participants) | 96 | 90
Percent change from baseline | -39.01 (13.04) | -40.07 (12.18)

3. Secondary Outcome: HDL-C
Description: Percent change from baseline in HDL-C level at Week 4
Time Frame: week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | 1PC002 | Lipitor
Number analyzed (Participants) | 96 | 90
Percent change from baseline | 0.06 (10.49) | -1.64 (11.01)

4. Secondary Outcome: Triglyceride
Description: Percent change from baseline in TG level at Week 4
Time Frame: week 4
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | 1PC002 | Lipitor
Number analyzed (Participants) | 96 | 90
Percent change from baseline | -18.75 (26.9) | -19.5 (25.5)

ADVERSE EVENTS:
Time Frame: 12-16 weeks
Groups:
- 1PC002: To summary the total adverse event of 1PC002.
- Lipitor: To summary the total adverse event of Lipitor.
Arm/Group | 1PC002 | Lipitor
Serious Adverse Events (participants affected / at risk) | 3/103 | 1/99
Other Adverse Events (participants affected / at risk) | 58/103 | 55/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1PC002 (N=103) | Lipitor (N=99)
Congestive heart failure (Cardiac disorders) | 0 | 1
Cellulitis,right hand (Infections and infestations) | 1 | 0
Rheumatic heart disease with Moderate Calcified Mitral stenosis (Cardiac disorders) | 1 | 0
Urinary tract infections (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1PC002 (N=103) | Lipitor (N=99)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Acute pulmonary oedema (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Lacrimation decreased (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 3 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Acute sinusitis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Pneumonia (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 9
Urinary tract infection (Infections and infestations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase (Investigations) | 9 | 6
Blood pressure increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 1
C-reactive protein abnormal (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
Hypotension (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 4
Sleep disorder (Psychiatric disorders) | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less